CLINICAL TRIAL: NCT05151497
Title: Effectiveness of Aquatic Theraphy in Spasticity: Watsu and Halliwick
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Miriam García Blanco, Principal investigator, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Universitiy of Cádiz
Record Dates: First submitted 2021-10-23; First posted 2021-12-09 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Brain-injury
Keywords: Acquired brain damage; aquatic therapy; hemiparesis; spasticity
MeSH Terms: conditions — Brain Injuries; Paresis; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Halliwick + Método Watsu (Experimental): The experimental group is made up of 7 subjects, the duration of the session being 75 minutes, divided into 45 minutes of Halliwick, 15 minutes of Watsu and finally 15 minutes of immersion in hot water. .
  In the application of the Halliwick Concept, it will be carried out in a pool at a temperature of 30ºC, and through the Ten Points Program.
  To carry out Watsu, the pool water must be at a temperature of 35ºC. The Watsu Basic Maneuver will be performed, consisting of a sequence of various positions where the subject must be as relaxed as possible, placed in a supine position, floating with eyes closed, and supported by the physiotherapist who is standing, with a wide base of support.
  Interventions: Other: Experimental group:Halliwick + Método Watsu
- Control group:Halliwick (Active Comparator): The control group is made up of 7 subjects, the duration of the session being 75 minutes, divided into 60 minutes of Halliwick and 15 minutes of immersion in hot water. Treatment using the Halliwick Concept is carried out in a pool where the water temperature is 30ºC, following the Ten Points Program.
  Interventions: Other: Control group:Halliwick

INTERVENTIONS:
Other: Experimental group:Halliwick + Método Watsu — Carrying out the Ten Points Program through the Halliwick Concept, together with the Watsu Method through a series of relaxation maneuvers and mobilization of the body in float, and an immersion time of 15 minutes without doing physical activity in a pool at a temperature of 30ºC , to decrease spasticity of various muscles.
  Arms: Experimental group: Halliwick + Método Watsu
Other: Control group:Halliwick — Exclusive use of treatment through the Halliwick Concept Ten Point Program, along with immersion in hot water to reduce spasticity in various muscles.
  Arms: Control group:Halliwick

SUMMARY:
Treatment with ACD patients will be carried out through the application of aquatic therapies, being the Halliwick Concept and the Watsu Method together with a time of immersion in hot water.

DETAILED DESCRIPTION:
The study consists of verifying the efficacy of physiotherapeutic treatment through the use of aquatic therapies, Watsu and Halliwick in subjects who have suffered Acquired Brain Injury (ACD), and who, after that, present spasticity. For this, the users of the Brain Injury Association of Cádiz (ADACCA) are taken as references.

Brain damage is a brain injury, resulting in a series of functional and neurological alterations. The treatment of this pathology will be carried out through the application of aquatic teràpies, being the Halliwick Concept and the Watsu Method.

This study consists of a clinical trial where the experimental group will be applied the combined treatment of Halliwick and Watsu together with a time of immersion in hot water, and to the control group the treatment by Halliwick plus immersion in hot water, in order to evaluate the degree of spasticity they present at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Belonging to the Acquired Brain Injury Association of Cádiz
* Presence of spasticity in the biceps brachii and soleus muscles confirmed by the modified Ashworth Scale and modified Tardieu Scale.
* Patients who are standing and walking at least with technical assistance and / or supervision.
* Patients with acquired brain damage and with spastic hemiparesis with a chronic evolution of more than 12 months.

Exclusion Criteria:

* Presence of infections.
* Other diagnosed diseases that prevent aquatic physiotherapy treatment, such as uncontrolled diabetes or dyspnea at rest.
* Have received aquatic therapy treatment in the six months prior to the study with the methods developed in the study (Halliwick or Watsu).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2021-12-27 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
Modified Asworth | Change from Baseline at 8 weeks
  0 (no increase in muscle tone) to 4 (rigid part in flex-ext)
  1 = Left
Modified Tardieu | Change from Baseline at 8 weeks
  0 (no resistance to movement) to 4 (10 second clonus)
Medical Outcome Study-Sleep Scale | Change from Baseline al 8 weeks
  Sleep rating (1 = more trouble falling asleep, a 6 = least trouble sleeping.
Number of years-Age | Baseline
  Years

CONTACTS AND LOCATIONS:
Overall Officials: Miriam García Blanco, Máster, Principal Investigator — University of Cadiz
Locations (3):
- Spain (3):
  - Miriam García Blanco, Cadiz, Cádiz
  - Asociación de Daño Cerebral de Cádiz (ADACCA), Cadiz, Cádiz
  - University of Cadiz, Cadiz